CLINICAL TRIAL: NCT02935972
Title: Pain Reduction During Transrectal Ultrasound-guided Biopsy of the Prostate: Intravenous Diazepam, Local Periprostatic Nerve Block or Combination
Brief Title: Combined Intravenous Diazepam, Local Periprostatic Nerve Block for Prostate Biopsy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MOHAMED F. MOSTAFA, lecturer of anesthesia and intensive care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Diazepam and TRUS Biopsy
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Pain Relief During Prostate Biopsy
Keywords: prostate biopsy, analgesia, anesthesia, pain, prostate cancer
MeSH Terms: conditions — Agnosia; Pain; Prostatic Neoplasms | interventions — Diazepam; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diazepam (Active Comparator): received intravenous diazepam 5 mg slowly just before TRUS probe insertion
  Interventions: Drug: Diazepam
- Local (Active Comparator): received 10 cc of 1% Lidocaine injected into the periprostatic nerve plexus bilaterally under ultrasound guidance
  Interventions: Drug: Lidocaine 1%
- Combined (Active Comparator): received intravenous diazepam 5 mg slowly just before TRUS probe insertion and 10 cc of 1% Lidocaine injected into the periprostatic nerve plexus bilaterally under ultrasound guidance
  Interventions: Drug: Diazepam and Lidocaine 1%

INTERVENTIONS:
Drug: Diazepam — received intravenous diazepam 5 mg slowly just before TRUS probe insertion
  Arms: Diazepam
Drug: Lidocaine 1% — received 10 cc of 1% Lidocaine injected into the periprostatic nerve plexus bilaterally under ultrasound guidance
  Arms: Local
Drug: Diazepam and Lidocaine 1% — received intravenous diazepam 5 mg slowly just before probe insertion and 10 cc of 1% Lidocaine injected into the periprostatic nerve plexus bilaterally under ultrasound guidance
  Arms: Combined

SUMMARY:
Prostate biopsy under transrectal ultrasound (TRUS) guidance is considered the procedure of choice for diagnosing prostate cancer. And as in any other diagnostic biopsy procedures; patients perceive anxiety before, during and after biopsy and ultrasound guided prostate biopsy is not an exclusion.

TRUS guided prostatic biopsies are mainly performed in an outpatient clinic, men undergoing transrectal prostate biopsy experience considerable psychological stress. It may be attributable to the fear of the potential diagnosis of cancer, the anal route of penetration, the fact that the subject organ examined is part of the sexual system and the anticipated pain and as a matter of fact the issues of discomfort and pain perceived throughout the procedure referred to the negative impact of the whole procedure, that is probe insertion and biopsy punctures.

Thus it is essential to employ a simple method that can liberate the patient from pain during prostate biopsy. Some studies recommend sedation , others recommend intra-rectal lidocaine gel and others periprostatic nerve block while others recommend Nitrous oxide inhalation as an effective method of analgesia for the procedural related pain or discomfort of prostate biopsy. The employment of analgesics, sedation and/or narcotic medication may alleviate much of the discomfort associated with transrectal prostate biopsy, such treatment may be associated with additional risks. Furthermore, when systemic medication is administered, patients require conscious sedation monitoring during and after the procedure, which may be inconvenient and relatively expensive in addition to their unsuitability to be performed on outpatient clinic basis. Therefore, a simple form of anesthesia is desirable.

Although a wide variety of anesthetic techniques are available for transrectal ultrasound-guided prostate biopsy, including rectal administration of lidocaine gel, periprostatic nerve blocks, intravenous propofol, and narcotic intramuscular premedication, these methods may not optimally prevent or relieve pain.

DETAILED DESCRIPTION:
From November 2013 to November 2014, 336 patients fitted our inclusion criteria underwent transrectal ultrasound-guided prostate biopsy (TRUSPB).

Informed consent was obtained from all patients after detail description of the study.

Bowel preparation with cleansing enema (a sodium phosphate and dibasic sodium phosphate enema) and antibiotic prophylaxis with Levofloxacin 500 mg. was prescribed.

Patients were randomized into three equal groups where Group I: to receive intravenous diazepam 5 mg slowly just before probe insertion Group II: received 10 cc of 1% Lidocaine injected into the periprostatic nerve plexus bilaterally under ultrasound guidance using a 22 gauge 7 inch needle , prior to injection caution was taken to aspirate before injection to avoid accidental intravascular injection of lidocaine, proper needle placement and injection of lidocaine a sonographic hypoechogenicity is created between the rectal wall and the base of the seminal vesicles causing the seminal vesicles to separate from the rectal wall and appear to be raised (fig.1) prostate biopsies had begun 2 to 3 minutes after lidocaine injection. Group III: intravenous diazepam 5 mg slowly just before probe insertion and 10 cc of 1% Lidocaine injected into the periprostatic nerve plexus bilaterally under ultrasound guidance.

Prostatic biopsies was performed in combined directed and random technique or extended random technique in absence of focal abnormality with mean number of biopsies 10 biopsies (9 to 12 biopsy) were done per patient.

The sedation scale were evaluated according to sedation scale. After the procedure, discomfort and pain experienced during performing the biopsy technique were graded using a 10-point linear visual analog pain scale.

All patients were monitored during and after the procedure for possible complications, patients were also questioned regarding any adverse effect at one week duration (at the time of receiving the histopathological results).

ELIGIBILITY:
Inclusion Criteria:

* abnormal digital rectal examination
* elevated PSA
* focal abnormality in TRUS.

Exclusion Criteria:

* previous allergy to diazepam or lidocaine
* bleeding diathesis or anticoagulant therapy
* history of chronic prostatitis
* acute anal and rectal conditions (as haemorrhoids, anal fissures or strictures)
* neurological conditions
* patients with respiratory asthma or chronic liver diseases

Ages: 40 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Score | 2 hours
  degree of pain during prostate biopsy

SECONDARY OUTCOMES:
Sedation Score | 2 hours
  degree of sedation during prostate biopsy
Complications | 2 hours
  hematuria, haematochezia or infection were recorded

CONTACTS AND LOCATIONS:
Overall Officials: HAMDY A. YOUSSEF, MD, Study Director — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided